CLINICAL TRIAL: NCT01614197
Title: A Phase I Trial of Temsirolimus (CCI-779, Pfizer, Inc.) in Combination With Etoposide and Cyclophosphamide in Children With Relapsed Acute Lymphoblastic Leukemia and Non-Hodgkins Lymphoma
Brief Title: A Trial of Temsirolimus With Etoposide and Cyclophosphamide in Children With Relapsed Acute Lymphoblastic Leukemia and Non-Hodgkins Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: T2014-001
Record Dates: First submitted 2012-05-18; First posted 2012-06-07 (Estimated); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Lymphoblastic Leukemia, Acute, Childhood; Lymphoblastic Lymphoma; Peripheral T-cell Lymphoma
Keywords: Relapse; Lymphoblastic; Leukemia; Refractory; Temsirolimus; Acute; Childhood; Pediatric; ALL; NHL; LL; PTL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Peripheral; Recurrence; Leukemia | interventions — temsirolimus; Etoposide; Cyclophosphamide; Methotrexate; Hydrocortisone; hydrocortisone hemisuccinate; Cytarabine

STUDY DESIGN:
Intervention Model Description: This study follows a standard 3+3 patient cohort escalation design, as described below:
  1. Three patients are entered at the first dose level
  2. If 0/3 experiences DLT at a given dose level, then the dose is escalated to the next higher level, if a higher dose level exists, and three patients are enrolled. If a higher dose level does not exists, up to three more patients are accrued at the same dose level.
  3. If 1/3 experiences DLT at current dose, then up to three more patients are accrued at the same dose level.
  4. If 2 or more DLTs are observed in a three-patient or six-patient cohort at a given dose level, then the MTD has been exceeded, dose escalation will be stopped, and up to three additional patients will be enrolled at the next lower dose level, if a lower dose level exists (unless six patients have already been treated at that prior dose).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level 1 (Experimental): This is the starting dose of temsirolimus at 7.5 mg/m^2 given IV. First dose of temsirolimus will be administered on Day 1, followed immediately by the first dose of IV etoposide and IV cyclophosphamide. Etoposide (100mg/m^2) and cyclophosphamide (440 mg/m^2) are continued for the next four days (Day 1-5). A second dose of temsirolimus is given on Day 8.
  Interventions: Drug: Temsirolimus; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Hydrocortisone; Drug: Cytarabine
- Dose Level 2 (Experimental): If Dose Level 1 is tolerated, the study will escalate to Dose Level 2 following the dose escalation schedule. Dose Level 2 will be administered via IV at 10 mg/m^2. First dose of temsirolimus will be administered on Day 1, followed immediately by the first dose of IV etoposide and IV cyclophosphamide. Etoposide (100mg/m^2) and cyclophosphamide (440 mg/m^2) are continued for the next four days (Day 1-5). A second dose of temsirolimus is given on Day 8.
  Interventions: Drug: Temsirolimus; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Hydrocortisone; Drug: Cytarabine
- Dose Level 3 (Experimental): If Dose Level 2 is tolerated, the study will escalate to Dose Level 3 following the dose escalation schedule. Dose Level 3 will be administered via IV at 15 mg/m^2. First dose of temsirolimus will be administered on Day 1, followed immediately by the first dose of IV etoposide and IV cyclophosphamide. Etoposide (100mg/m^2) and cyclophosphamide (440 mg/m^2) are continued for the next four days (Day 1-5). A second dose of temsirolimus is given on Day 8.
  Interventions: Drug: Temsirolimus; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Hydrocortisone; Drug: Cytarabine
- Dose Level 4 (Experimental): If Dose Level 3 is tolerated, the study will escalate to Dose Level 4 following the dose escalation schedule. Dose Level 4 will be administered via IV at 25 mg/m^2. First dose of temsirolimus will be administered on Day 1, followed immediately by the first dose of IV etoposide and IV cyclophosphamide. Etoposide (100mg/m^2) and cyclophosphamide (440 mg/m^2) are continued for the next four days (Day 1-5). A second dose of temsirolimus is given on Day 8. Temsirolimus will not be escalated beyond Dose Level 4.
  Interventions: Drug: Temsirolimus; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Hydrocortisone; Drug: Cytarabine

INTERVENTIONS:
Drug: Temsirolimus — Dose will be assigned at study entry. Give IV over 30 minutes on days 1 and 8.
  Other Names: Torisel; CCI-779
Drug: Etoposide — 100 mg/m2 IV over 1-2 hours daily x 5 on Days 1-5.
  Other Names: Toposar; VePesid; VP-16
Drug: Cyclophosphamide — 440 mg/m2 IV daily x 5 on Days 1-5 given over 30-60 minutes.
  Other Names: Cytoxan; Neosar
Drug: Methotrexate — PATIENTS WITH CNS 1 COURSES 2, 4, 6, 8: Give intrathecally to patients who were CNS1 at study entry day 1 of each course at the doses listed below.
  * Age 1 - 1.99 give 8 mg of methotrexate
  * Age 2 - 2.99 give10 mg of methotrexate
  * Age 3 - 8.99 give 12 mg of methotrexate
  * Age ≥ 9 give 15 mg of methotrexate
  PATIENTS WITH CNS 2 or 3 DISEASE
  -COURSE 1: Give intrathecally to patients with CNS 2 or 3 disease at the doses defined by age below on day 6 and then weekly until the patient is CNS 1.
  COURSES 2-8: Give intrathecally to patients who were CNS 3 at study entry on day 1 of each course.
  * 8 mg for patients age 1-1.99
  * 10 mg for patients age 2-2.99
  * 12 mg for patients 3-8.99 years of age
  * 15 mg for patients >9 years of age
  Other Names: MTX; Amethopterin; Trexall
Drug: Hydrocortisone — Given with Methotrexate and Cytarabine for patients with CNS 2 or 3 disease.
  COURSE 1: Give intrathecally to patients with CNS 2 or 3 disease at the doses defined by age below on day 6 and then weekly until the patient is CNS 1.
  COURSES 2-8: Give intrathecally to patients who were CNS 3 at study entry on day 1 of each course.
  * 8 mg for patients age 1-1.99
  * 10 mg for patients age 2-2.99
  * 12 mg for patients 3-8.99 years of age
  * 15 mg for patients >9 years of age
  Other Names: Hydrocortisone sodium succinate; Solu-cortef
Drug: Cytarabine — For Patients who are CNS1 COURSE 1: Give intrathecally to patients with CNS1 disease at the dose defined by age below on day 1 of course 1 if no other IT was given within 1 week of day 1 of course 1
  * Age 1 - 1.99 give 30 mg of Cytarabine
  * Age 2 - 2.99 give 50mg of Cytarabine
  * Age ≥ 3 give 70 mg of Cytabine
  For Patients with CNS 2 or 3 Disease COURSE 1: Give intrathecally to patients with CNS 2 or 3 disease at the doses defined by age below on day 1 if no other IT chemotherapy given within 1 week of day 1 of course 1. Then give weekly until the patient is CNS 1 or 2 (investigator discretion). No more than 5 weekly doses to be given in cycle 1.
  COURSES 2-8: Give intrathecally to patients who were CNS 2or 3 at study entry on day 1 of each course.
  * 16 mg for patients age 1-1.99
  * 20 mg for patients age 2-2.99
  * 24 mg for patients 3-8.99 years of age
  * 30 mg for patients >9 years of age
  Other Names: Cytosine arabinoside; Ara-C; Cytosar

SUMMARY:
This is a phase I study of temsirolimus (Torisel) combined with dexamethasone, cyclophosphamide and etoposide in patients with relapsed acute lymphoblastic leukemia (ALL), lymphoblastic lymphoma (LL) or peripheral T-cell lymphoma (PTL).

DETAILED DESCRIPTION:
Studies have shown that mTOR inhibitors (MTI) inhibit growth of pre-B and T-cell ALL cell lines in vitro and in ALL xenograft models. The MTI temsirolimus was chosen for use in this study due to its weekly intravenous dosing, its more predictable blood levels, and availability of a single-agent pediatric MTD and its sustained biologic effect due to conversion to sirolimus. This study will determine the maximum tolerated dose of temsirolimus that can given in combination with dexamethasone, cyclophosphamide and etoposide in relapsed ALL, LL or PTL. A standard 3-patient cohort dose-escalation design will be used. Response to treatment will be evaluated. Biology tests will be done to evaluate minimal residual disease (MRD), temsirolimus' effect on glucocorticoid resistance, and mTOR inhibition.

ELIGIBILITY:
INCLUSION CRITERIA

-Patients must be greater than or equal to 12 months and ≤ 21 years of age at the time of study enrollment.

Patients must have one of the following:

Leukemia

* Bone marrow involvement defined as ALL ≥ 25% blasts (M2 or M3) with or without extramedullary involvement.
* Refractory bone marrow involvement defined as MRD ≥ 0.1% blasts done at a COG-approved MRD testing lab after most recent treatment regimen. in the bone marrow (M23) and any CNS status. OR
* Newly diagnosed patients (T or B-cell ALL) with refractory bone marrow involvement after Consolidation therapy are eligible.
* First relapse B-cell ALL patients are eligible with refractory disease.
* Second or greater relapse B-cell patients are eligible at time of relapse or with refractory disease.
* First or greater relapse T-cell ALL patients are eligible at time of relapse or with refractory disease.
* Isolated CNS 2 or 3 patients with < 0.1% MRD bone marrow involvement are not eligible.

Lymphoma

* Patient must have relapsed or refractory lymphoblastic lymphoma or peripheral T-cell lymphoma.
* Patient must have histologic verification of disease at original diagnosis.
* Patient must have evaluable or measurable disease documented by clinical or radiographic criteria or bone marrow disease present at study entry.
* Patients may have CNS 2 or 3 disease

Karnofsky greater than or equal to 50% for patients > 16 years of age and Lansky greater than or equal to 50 for patients ≤ 16 years of age.

Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy.

Patients with leukemia or lymphoma who relapse while receiving maintenance chemotherapy will not be required to have a waiting period before enrollment onto this study.

At least 14 days must have elapsed after the completion of cytotoxic therapy, with the exception of hydroxyurea.

Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor.

Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair

Immunotherapy: At least 30 days after the completion of any type of immunotherapy, e.g. tumor vaccines. or chimeric antigen receptor T cell (CART) therapy or tumor vaccines.

Monoclonal antibodies: At least 3 half-lives of the antibody must have elapsed after the last dose of a monoclonal antibody. (ie: Rituximab = 66 days, Epratuzumab = 69 days). Patients must have been off blinatumomab infusion for at least 4 days and all drug-related toxicity must have resolved to grade 2 or lower as outlined in the inclusion and exclusion criteria

XRT: At least 14 days after local palliative XRT (small port); At least 84 days must have elapsed if prior TBI, craniospinal XRT or if greater than or equal to 50% radiation of pelvis; At least 42 days must have elapsed if other substantial marrow radiation.

Stem Cell Infusion: No evidence of active graft vs. host disease and at least 84 days must have elapsed after transplant or stem cell infusion.

Adequate Bone Marrow Function Defined as: Blood counts are not required to be normal prior to enrollment on trial. However, platelet count must be greater than or equal to 20,000/mm3 to initiate therapy (may receive platelet transfusions). Patients should not be known to be refractory to red blood cell or platelet transfusions.

Adequate Renal Function Defined as:

* Creatinine clearance or radioisotope GFR greater than or equal to 70ml/min/1.73 m2 or
* Normal serum creatinine based on age and gender.

Adequate Liver Function Defined as:

* Total bilirubin (sum of conjugated + unconjugated) must be less than or equal to 1.5 x normal per institutional normal values for age.
* SGPT (ALT) and SGOT (AST) must be less than 3 x institutional upper limit of normal (Grade 1 or less per CTCAE 4).

  --GGT must be less than 2.5 x institutional upper limit of normal (Grade 1 or less per CTCAE 4).
* Serum albumin greater than or equal to 2 g/dL.
* The hepatic requirements may be waived for patients with elevations clearly due to leukemic infiltration after consultation with the Study Chair or Vice Chair.
* Fasting or non-fasting serum triglyceride level ≤ 300 mg/dL and serum cholesterol level ≤ 300 mg/dL.

Adequate Cardiac Function Defined As:

* Shortening fraction of ≥ 27% by echocardiogram, or
* Ejection fraction of ≥ 50% by gated radionuclide study.

Adequate Pulmonary Function Defined as:

* Pulse oximetry > 94% on room air (> 90% if at high altitude)
* No evidence of dyspnea at rest and no exercise intolerance.
* Baseline chest x-ray with no evidence of active infectious disease or pneumonitis.

Reproductive Function

* Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed prior to enrollment.
* Female patients with infants must agree not to breastfeed their infants while on this study.
* Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study.
* Random or fasting glucose within the upper limits of normal for age. If the initial blood glucose is non-fasting and above normal limits a fasting glucose can be obtained and must be within the upper limits of normal for age.

EXCLUSION CRITERIA

* Corticosteroids: Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible.
* Investigational Drugs: Patients who are currently receiving another investigational drug are not eligible. The definition of "investigational" for use in this protocol means any drug that is not licensed by the FDA, Health Canada or the Therapeutic Goods Administration to be sold in the countries they govern. (United States, Canada and Australia)
* Anti-cancer Agents: Patients who are currently receiving or may receive while on therapy, other anti-cancer agents, radiation therapy or immunotherapy are not eligible [except leukemia patients receiving hydroxyurea, which may be continued until 24 hours prior to start of protocol therapy]. Intrathecal chemotherapy (at the discretion of the primary oncologist) may be given up to one week prior to the initiation of study therapy.
* Anti-GVHD or agents to prevent organ rejection post-transplant: Patients who are receiving cyclosporine, tacrolimus or other agents to prevent either graft-versus-host disease post bone marrow transplant or organ rejection post transplant are not eligible for this trial. At least 3 half-lives must have elapsed after the last dose of GVHD meds.
* Anticoagulants: Patients who are currently receiving therapeutic anticoagulants (including aspirin, low molecular weight heparin, and others) are not eligible. At least 3 half-lives must have elapsed after the last dose of anticoagulants.
* Angiotensin-converting enzyme (ACE) inhibitors: Patients who are currently receiving ACE inhibitors are not eligible due to the development of angioneurotic edema-type reactions in some subjects who received concurrent treatment with temsirolimus + ACE inhibitors. At least 3 half-lives must have elapsed after the last dose of ACE inhibitors.
* Calcium Channel Blockers: Patients who are currently receiving Calcium Channel Blockers are not eligible due to the development of angioneurotic edema-type reactions in some subjects who received concurrent treatment with temsirolimus + Calcium Channel Blockers. At least 3 half-lives must have elapsed after the last dose of Calcium Channel Blockers.
* Enzyme inducing Anti-convulsants: Patients who are currently receiving enzyme inducing anticonvulsants (ie phenytoin, phenobarbitol, or carbamazepine) are not eligible. Stabilizing on a non-hepatic inducing metabolizing anti-convulsant (ie: gabapentin or levetiracetam) prior to study entry is acceptable. At least 3 half-lives must have elapsed after the last dose of enzyme inducing anti-coagulants.
* Patients receiving treatment with azoles such as fluconazole or voriconazole which are potent inhibitors of temsirolimus metabolism. At least 3 half-lives must have elapsed after the last dose of azoles.
* Patient with Burkiett's leukemia and /or lymphoma are not eligible.

Infection Criteria

Patients are excluded if they have:

* Positive blood culture within 48 hours of study enrollment;
* Fever above 38.2 within 48 hours of study enrollment with clinical signs of infection. Fever that is determined to be due to tumor burden is allowed if patients have documented negative blood cultures for at least 48 hours prior to enrollment and no concurrent signs or symptoms of active infection or hemodynamic instability.
* A positive fungal culture within 30 days.
* Active fungal, viral, bacterial, or protozoal infection requiring IV treatment. Chronic prophylaxis therapy to prevent infections is allowed.

Patients with Down syndrome and Fanconi Anemia are excluded.

Patients will be excluded if they have significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance with protocol treatment or required observations, interfere with consent, study participation, follow up, or interpretation of study results.

Patients with known optic nerve and/or retinal involvement (because it may not be possible to safely delay irradiation) are not eligible. Patients presenting with visual disturbances by history or physical exam should have an ophthalmological exam and, if indicated, an MRI to determine optic nerve or retinal involvement.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2015-07-03 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Rheingold, MD, Study Chair — Children's Hospital of Philadelphia
Locations (32):
- United States (25):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Orange County, Orange, California
  - UCSF School of Medicine, San Francisco, California
  - The Children's Hospital, University of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami Cancer Center, Miami, Florida
  - Children's Healthcare of Atlanta, Emory University, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Childrens Hospital & Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Hospital New York-Presbyterian, New York, New York
  - Levine Children's Hospital at Carolinas Medical Center, Charlotte, North Carolina
  - Rainbow Babies, Cleveland, Ohio
  - Nationwide Childrens Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude, Memphis, Tennessee
  - University of Texas at Southwestern, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Royal Children's Hospital, Melbourne, Melbourne, Victoria
  - Sydney Children's Hospital, Sydney
- Canada (3):
  - Hospital for Sick Kids, Toronto, Ontario
  - Sainte Justine University Hospital, Montreal, Quebec
  - British Columbia Children's Hospital, Vancouver

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: This is the starting dose of temsirolimus at 7.5 mg/m^2 given IV. First dose of temsirolimus will be administered on Day 1, followed immediately by the first dose of IV etoposide and IV cyclophosphamide. Etoposide and cyclophosphamide are continued for the next four days (Day 1-5). A second dose of temsirolimus is given on Day 8.
  Temsirolimus: Dose will be assigned at study entry. Give IV over 30 minutes on days 1 and 8.
  Etoposide: 100 mg/m2 IV over 1-2 hours daily x 5 on Days 1-5.
  Cyclophosphamide: 440 mg/m2 IV daily x 5 on Days 1-5 given over 30-60 minutes.
- Dose Level 2: If Dose Level 1 is tolerated, the study will escalate to Dose Level 2 following the dose escalation schedule. Dose Level 2 will be administered via IV at 10 mg/m^2. First dose of temsirolimus will be administered on Day 1, followed immediately by the first dose of IV etoposide and IV cyclophosphamide. Etoposide and cyclophosphamide are continued for the next four days (Day 1-5). A second dose of temsirolimus is given on Day 8.
  Temsirolimus: Dose will be assigned at study entry. Give IV over 30 minutes on days 1 and 8.
  Etoposide: 100 mg/m2 IV over 1-2 hours daily x 5 on Days 1-5.
  Cyclophosphamide: 440 mg/m2 IV daily x 5 on Days 1-5 given over 30-60 minutes.
- Dose Level 3: If Dose Level 2 is tolerated, the study will escalate to Dose Level 3 following the dose escalation schedule. Dose Level 3 will be administered via IV at 15 mg/m^2. First dose of temsirolimus will be administered on Day 1, followed immediately by the first dose of IV etoposide and IV cyclophosphamide. Etoposide and cyclophosphamide are continued for the next four days (Day 1-5). A second dose of temsirolimus is given on Day 8.
  Temsirolimus: Dose will be assigned at study entry. Give IV over 30 minutes on days 1 and 8.
  Etoposide: 100 mg/m2 IV over 1-2 hours daily x 5 on Days 1-5.
  Cyclophosphamide: 440 mg/m2 IV daily x 5 on Days 1-5 given over 30-60 minutes.
- Dose Level 4: If Dose Level 3 is tolerated, the study will escalate to Dose Level 4 following the dose escalation schedule. Dose Level 4 will be administered via IV at 25 mg/m^2. First dose of temsirolimus will be administered on Day 1, followed immediately by the first dose of IV etoposide and IV cyclophosphamide. Etoposide and cyclophosphamide are continued for the next four days (Day 1-5). A second dose of temsirolimus is given on Day 8. Temsirolimus will not be escalated beyond Dose Level 4.
  Temsirolimus: Dose will be assigned at study entry. Give IV over 30 minutes on days 1 and 8.
  Etoposide: 100 mg/m2 IV over 1-2 hours daily x 5 on Days 1-5.
  Cyclophosphamide: 440 mg/m2 IV daily x 5 on Days 1-5 given over 30-60 minutes.
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Started | 3 | 4 | 6 | 3
Completed | 3 | 3 | 6 | 3
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of patients who were enrolled onto the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Total
Number analyzed (Participants) | 3 | 4 | 6 | 3 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 6 | 3 | 16
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 4 | 2 | 6
  Male | 3 | 4 | 2 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 6 | 1 | 8
  Not Hispanic or Latino | 2 | 3 | 0 | 2 | 7
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 3 | 3 | 3 | 1 | 10
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 1 | 0 | 0 | 2
  United States | 2 | 3 | 6 | 2 | 13
  Australia | 0 | 0 | 0 | 1 | 1
Prior Therapy Regimens [Count of Participants; unit: Participants] — Population: Total number of patients that were enrolled onto the study
  Participants
    # of prior therapies : 1 prior therapy | 0 | 0 | 0 | 0 | 0
    # of prior therapies : 2 prior therapies | 0 | 1 | 1 | 1 | 3
    # of prior therapies : 3 prior therapies | 2 | 1 | 2 | 0 | 5
    # of prior therapies : 4 prior therapies | 0 | 0 | 0 | 0 | 0
    # of prior therapies : 5 prior therapies | 0 | 1 | 1 | 2 | 4
    # of prior therapies : 6 prior therapies | 0 | 0 | 0 | 0 | 0
    # of prior therapies : 7 prior therapies | 1 | 0 | 2 | 0 | 3
    Prior transplant : Yes | 2 | 2 | 4 | 0 | 8
    Prior transplant : No | 1 | 1 | 2 | 3 | 7
    Prior CAR-T cell therapy : Yes | 1 | 0 | 2 | 1 | 4
    Prior CAR-T cell therapy : No | 2 | 3 | 4 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Experienced DLT During Cycle 1 of Therapy
Description: The incidence of dose limiting toxicity (DLT) will be measured. The maximum tolerated dose will be the highest study dose at which 1 or fewer of six patients experience DLT during cycle 1 of therapy. All these analyses will be descriptive and exploratory and hypotheses generating in nature.
Time Frame: Cycle 1 (a minimum of 4 weeks and a max of 8 weeks)
Population: Number of patients that initiated and completed study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 3 | 3 | 6 | 3
Participants
  Number of patients that did not experience DLT | 3 | 3 | 5 | 3
  Number of patient that did experience DLT | 0 | 0 | 1 | 0

2. Secondary Outcome: Response Rate at the Completion of 1 Cycle of Study Treatment
Description: CR = Complete remission defined as attainment of bone marrow with <5% blasts with no evidence of circulating blasts or extramedullary disease and with recovery of peripheral counts (absolute neutrophil counts (ANC) > or = to 500/uL and platelet count > or = to 50,000 microliters) CRi = Complete remission with incomplete blood count recovery defined as attainment of bone marrow with >5% blasts with no evidence of circulating blasts or extramedullary disease but insufficient recovery of ANC < 500/uL or platelets < 50,000 microliters PR = partial remission defined as complete disappearance of circulating blasts and achievement of 5-25% blasts if greater than 25% blasts originally without new sites of extramedullary disease and with recovery of ANC.
  SD = stable disease defined as not satisfying criteria for PD, or has recovery of ANC > or = to 500/uL and fails to qualify for CR, CRi, or PR PD = progressive disease defined as an increase of at least 25% in bone marrow leukemic cells
Time Frame: Cycle 1 (a minimum of 4 weeks and a max of 8 weeks)
Population: All these analyses will be descriptive and exploratory and hypotheses generating in nature.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 3 | 3 | 6 | 3
Participants
  CR | 0 | 1 | 1 | 0
  CRi | 1 | 0 | 0 | 1
  PR | 1 | 1 | 1 | 0
  SD | 0 | 1 | 1 | 1
  PD | 1 | 0 | 3 | 1

3. Secondary Outcome: Minimum Residual Disease (MRD) Levels Present at End of Cycle 1 Therapy in Patients
Description: MRD positive is defined as > or = to 0.1% MRD MRD negative is define as < 0.1% MRD
  All these analyses will be descriptive and exploratory and hypotheses generating in nature.
Time Frame: Cycle 1 (a minimum of 4 weeks and a max of 8 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 3 | 3 | 6 | 3
Participants
  MRD positive | 3 | 2 | 5 | 2
  MRD negative | 0 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to 60 days
Description: The definition of adverse event and/or serious adverse event used to collect adverse event information is the same as clinicaltrials.gov.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
All-Cause Mortality (participants affected / at risk) | 3/3 | 1/3 | 3/6 | 2/3
Serious Adverse Events (participants affected / at risk) | 3/3 | 0/3 | 3/6 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=6) | Dose Level 4 (N=3)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=6) | Dose Level 4 (N=3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 5 (5) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 5 (5) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 5 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bicarbonate serum low (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased respiratory rate (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diaper rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 1 (1) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dystonic reaction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ear skin cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated creatinine (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated lactic acid (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infection (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Erythematous rash (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 3 (3) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (3) | 2 (2) | 3 (3) | 1 (1)
GGT increased (Investigations) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (5) | 1 (1) | 2 (3) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Hypochloremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0) | 4 (4) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 5 (5) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 3 (5) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased respiratory rate (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Klebsiella oxytoca (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 3 (3) | 3 (3) | 0 (0)
Marked osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 2 (2) | 5 (5) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (5) | 2 (2) | 4 (6) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3) | 2 (2) | 5 (5) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital edema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perirectal erythema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perirectal excoriation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 2 (2) | 5 (5) | 3 (3)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Pseudomonas aeruginosa in blood (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PTT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcus epidermidis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Urine output decreased (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 3 (3) | 3 (3) | 5 (5) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
All these analyses will be descriptive and exploratory and hypotheses generating in nature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT01614197/Prot_SAP_000.pdf